CLINICAL TRIAL: NCT05175989
Title: Real-world SARS-CoV-2 Antibody Response in Children Aged 5-11 Years Following BNT162b2 mRNA Vaccination Against COVID-19: a Prospective Cohort Study
Brief Title: SARS-CoV-2 Antibody Response in Children Aged 5-11 Years Following Vaccination Against COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0810-21-RMC
Record Dates: First submitted 2021-12-30; First posted 2022-01-04 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are few data on the immunogenicity of the Pfizer-Biontec BNT162b2 vaccine for the prevention of COVID-19 disease and of side effects in children aged 5-11 years. Therefore, our aim is to determine the immunogenicity and to describe the local or systemic reactogenicity events after vaccination with the BNT162b2 COVID-19 vaccine in children aged 5-11 years for a period of six and half months following the first dose of the vaccine.

DETAILED DESCRIPTION:
The Pfizer-Biontec BNT162b2 vaccine has proven efficacy and safety for the prevention of COVID-19 disease in adults and adolescents aged 12 years and older. Efficacy and safety were recently shown also for children aged 5-11 years. Side-effects are common, including some rare but important side-effects such as myocarditis. Myocarditis post Pfizer-Biontec BNT162b2 vaccination was described mostly among male adolescents and young adults. There are few data on the immunogenicity of the vaccine and of side effects in children aged 5-11 years. Therefore, our aim is to determine the immunogenicity and to describe the local or systemic reactogenicity events after vaccination with the BNT162b2 COVID-19 vaccine in children aged 5-11 years.

This is a prospective cohort study assessing the immunogenicity of the BNT162b2 COVID-19 vaccine in children. The study population will be composed of children aged 5-11 years at the Schneider Children's Medical Center, with no contraindication for COVID-19 vaccination. Upon enrollment in the study, participates will be requested to complete an enrollment questionnaire and a blood sample for baseline serological evaluation will be obtained.

The study follow-up period will be 6 and a half months from receipt of the first dose of the vaccine. The study will last 6 months from the date of the approval of the study protocol.

Blood samples for immune response evaluation will be taken at intervals of 28 days (+/- 14) until 6 and a half months from receipt of the first dose of the vaccine. Samples will be tested for antibodies to SARS-CoV-2 at the Microbiology Laboratory at the Rabin Medical Center. Symptomatic participants with any respiratory symptoms or other symptoms suggestive of COVID-19 disease will be tested for SARS-CoV-2 by RT-PCR, at laboratories certified by the Ministry of Health.

ELIGIBILITY:
Inclusion Criteria:

Age 5-11 years

Exclusion Criteria:

Administration of COVID-19 vaccine>21 days prior to enrollment, Contraindication for COVID-19 vaccine such as, known hypersensitivity to a component of the vaccine or its excipients Congenital or acquired immunodeficiency (including recipient of systemic steroids ≥2 mg/kg or ≥20mg/day, within two weeks prior to enrollment)

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 5-11 years eligible for BNT162b2 vaccine
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of the Pfizer-Biontec BNT162b2 COVID-19 vaccine in children aged 5-11 years. Our second aim is to describe the local or systemic reactogenicity events after vaccination with the BNT162b2 COVID-19 vaccine in children | Day 56 (day 43 to 70) (28 days +/- 14 days after second injection)
  SARS-CoV-2 serum antibody levels

SECONDARY OUTCOMES:
local or systemic reactogenicity events after vaccination with the BNT162b2 COVID-19 vaccine in children aged 5-11 years | Up to Day 56 (day 43 to 70) (28 days +/- 14 days after second injection)
  Description of side effects
Evaluation of the long-term immune response following the BNT162b2 vaccine by SARS-CoV-2 serum antibody levels that meet or exceed the threshold of protection From COVID-19 | Day 84 (71-98), day 112 (99-126), day 140 (127-154), day 168 (155-182), day 196 (183-197)].
  long-term immune response
Seroresponse rate of vaccine recipients (greater than or equal to 4-fold rise from before vaccination in SARS-CoV-2 serum antibody levels | Day 56 (day 43 to 70) (28 days +/- 14 days after second injection)
  Seroresponse rate
Number of participants with medically-attended AEs (MAAEs) | Up to Day 56 ((day 43 to 70) (28 days +/- 14 days after second injection)
  medically-attended AEs
Number of participants with serious adverse events (SAEs) | Up to Day 56 ((day 43 to 70) (28 days +/- 14 days after second injection)
  erious adverse events (SAEs)
Number of Participants with Adverse Events of Special Interest (AESIs), Including Multisystem Inflammatory Syndrome in Children (MIS-C) | Up to Day 56 (day 43 to 70) (28 days +/- 14 days after second injection)
  Adverse Events of Special Interest (AESIs)

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No